CLINICAL TRIAL: NCT00350038
Title: Investigations of the Effects of Aprovel, Lipanor and Their Combination Onto the Endothelial Functions of Dyslipidemic Patients Measure by Laser Doppler Flow-Metry.
Brief Title: Irbesartan, Ciprofibrate and Their Combination Onto the Endothelial Functions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L_8759
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Irbesartan; ciprofibrate

INTERVENTIONS:
Drug: Irbesartan
Drug: Ciprofibrate

SUMMARY:
The rationale of the study is to clarify whether the supplementation of irbesartan with ciprofibrate could increase the antihypertensive effect, could improve the endothelial functions, and/or could affect the atherogenic small-dense LDL-, oxydized LDL concentrations, onto the paraoxinase activity and on the CRP and insulin levels.

ELIGIBILITY:
Inclusion Criteria:

* hypertensive + dyslipidemic + damaged endothelial function

Exclusion Criteria:

* hepatic and kidney damage,
* IDDM (Insulin Dependent Diabetes Mellitus)
* Freckson V type hyperlipoproteinaemia

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-02; Study Completion 2007-08

PRIMARY OUTCOMES:
Microvascular reactivity

SECONDARY OUTCOMES:
Reach of target blood pressure
Measurements of safety laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: László Erős, MD, Study Director — Sanofi-aventis, Hungary
Locations (1):
- Sanofi-aventis, Budapest, Hungary